CLINICAL TRIAL: NCT03515356
Title: Exercise to Reduce Chemotherapy-Induced Peripheral Neuropathy: A Pilot RCT
Brief Title: Exercise to Reduce Chemotherapy-Induced Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2018.023; HUM00136639 (Other: University of Michigan)
Record Dates: First submitted 2018-04-22; First posted 2018-05-03 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Gastrointestinal Cancer; Colorectal Cancer; Pancreatic Cancer; Gastric Cancer; Stomach Cancer; Esophageal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MI-Walk Intervention (Experimental): Subjects who are already receiving oxaliplatin prescribed by their oncologist (as standard of care) will receive a physical activity education pamphlet.
  In addition, subjects will receive 8-weeks of motivational enhancement therapy- and a home-based aerobic walking intervention. Motivational interviewing will be delivered with concurrent feedback and motivational techniques in 30-45-minute sessions at intervention orientation (T1), 2 weeks (T3), and 4 weeks (T4).
  Interventions: Behavioral: MI-Walk Intervention; Behavioral: Physical Activity Education Pamphlet
- PA Education Alone (Active Comparator): Subjects who are already receiving oxaliplatin prescribed by their oncologist (as standard of care) will receive a physical activity education pamphlet.
  Interventions: Behavioral: Physical Activity Education Pamphlet

INTERVENTIONS:
Behavioral: MI-Walk Intervention — Eight-week motivational enhancement therapy and home-based aerobic walking intervention
  Arms: MI-Walk Intervention
Behavioral: Physical Activity Education Pamphlet — Physical activity education pamphlet only

SUMMARY:
This randomized, controlled, pilot experiment will evaluate the effects of an aerobic walking intervention on OIPN (oxaliplatin-induced peripheral neuropathy) in patients with gastrointestinal (GI) cancer who are already prescribed oxaliplatin (85 mg/m2 every other week for at least six cycles) by their oncologists. Oxaliplatin is a standard chemotherapy treatment for invasive GI cancers that causes OIPN in 85-95% of patients.

DETAILED DESCRIPTION:
Background: Over 190,000 men and women will be diagnosed in 2018 with invasive gastrointestinal (GI) cancers (e.g, colorectal and gastric cancer) for which oxaliplatin is a standard chemotherapy treatment. However, 85-95% of these patients develop oxaliplatin-induced peripheral neuropathy (OIPN). Currently, OIPN is the primary dose-limiting factor of oxaliplatin-based regimens, because persistent OIPN can impair physical function and quality of life (QOL) years after treatment completion. There are no effective treatments for OIPN. Four randomized controlled trials and two quasi-experiments have reported positive effects of at least 10 minutes/day of moderate-intensity aerobic exercise, 2-5 days/week over at least 6-8 weeks on chemotherapy-induced peripheral neuropathy. Exercise-enhanced circulation could re-distribute neurotoxic drugs away from vulnerable neurons, reduce oxidative stress, and help to prevent OIPN. However, all the prior trials had critical study limitations and all but two studies evaluated OIPN as a secondary outcome. Thus, this prospective, randomized, controlled, pilot experiment will evaluate the efficacy of an aerobic walking intervention for OIPN in GI cancer patients who are already prescribed oxaliplatin (85 mg/m2 every other week for at least six cycles) by their oncologists. The "MI-Walk intervention"- an 8-week motivational enhancement therapy (MET)- and home-based aerobic walking intervention-will be tested in this study.

Specific aims: The specific aims and hypotheses are to:

Aim 1: Evaluate the effect of the MI-Walk Intervention on OIPN severity at 8 weeks (T6) compared to physical activity (PA) education alone.

Hypothesis: Participants who receive the MI-Walk intervention will exhibit less severe OIPN at T6 than participants who receive PA education alone.

Aim 2: Explore the effect of the MI-Walk intervention on total oxaliplatin received, and QOL at T6 compared to PA education alone.

Hypothesis: Participants who receive the MI-Walk intervention will receive higher total doses of oxaliplatin and report higher QOL at T6 than participants who receive PA education alone.

Aim 3: Evaluate the feasibility of the MI-Walk intervention. Research Questions: Among patients receiving oxaliplatin, 1) how acceptable is the intervention? 2) what percent of patients will enroll in, complete, and adhere to the walking intervention? 3) what participant characteristics are associated with study compliance, adherence, completion, and acceptability? 4) What, if any, adverse events will result from the MI-Walk intervention?

Study design: Sixty GI cancer patients will be recruited at multiple cancer clinics within the week before their second oxaliplatin cycle. All participants will receive a PA education pamphlet. Half (n=30) will receive the MI-Walk Intervention. These patients will receive a tailored progressive walking plan, supplemental cancer treatment & exercise education, patient testimony, HR-enabled pedometer and PA-tracking app, exercise diary, and semi-scripted brief MET (motivational interviewing, SMAART goals, and if-then statements) from research staff before practicing the intervention at home for 8 weeks. Additional brief MET sessions at 2 (T3) and 4 weeks (T4), progress summaries at T3, T4, and T6, a private email group, weekly group walking events, and peer accountability phone calls/email will be used to engage and support participants. To level attention, both groups will receive regular phone assessments of intervention-related adverse events at 1 week (T2), T3, T4, and 6 weeks (T5). Outcomes will be measured at (T1) and 8 weeks after (T6) intervention initiation. The outcome measures include the 0-10 NRS of OIPN symptom severity (primary outcome measure); and EORTC QLQ-CIPN20 self-report survey, cumulative oxaliplatin dose, and EORTC QLQ-C30. The study will also record feasibility, adherence, acceptability, and intervention fidelity data. Multiple linear regression will be used to evaluate the inter-group differences in the T1 to T6 change in mean NRS scores (OIPNΔ), controlling for T6 total oxaliplatin received (OXALIT6), and the interaction between the intervention and OXALIT6. Mediation analysis will be used to explore the secondary outcomes.

Future Directions: This study will be among the first to provide efficacy and feasibility data for an 8-week home-based aerobic walking intervention to reduce OIPN - a common chemotherapy side effect, for which there are no good treatments. This pilot study will inform the design of larger phase III trials to evaluate the efficacy of aerobic walking for OIPN, and potential mediators (e.g., vascular biomarkers) in this relationship.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed GI cancer (e.g, colorectal, gastric, pancreatic, esophageal, bowel);
* Scheduled to receive at least 6 cycles of oxaliplatin (85 mg/m2);
* Receiving care at the University of Michigan or St. Joseph Cancer Clinics;
* A Karnofsky Performance Status ≥ 80% or an Eastern Cooperative Oncology Group Status 0 to 1;
* Voluntarily consented to participate in all intervention components.

Exclusion Criteria:

* Exercise- or mobility-limiting cardiovascular, pulmonary, musculoskeletal, or psychological disease, based on the EMR (electronic medical record) past medical history and consultation with the medical oncologist;
* Scheduled major surgery during the study time period;
* Pre-existing peripheral neuropathy prior to chemotherapy (potentially due to diabetes, central nervous system malignancy, vitamin deficiency, heredity, nerve compression injury, non-surgically corrected carpal tunnel disease, or alcohol dependence) per patient self-report in response to brief screening questions noted in the pre-screening section;
* Pregnancy;
* Inability to read or speak English;
* Prognosis of less than three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Sensory neuropathy at 8 weeks | At 8 weeks
  The 9-item European Organisation of Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-Chemotherapy-Induced Peripheral Neuropathy Scale (CIPN20) sensory subscale will be used to measure sensory neuropathy. Each item is rated on a scale from 1 ("not at all") to 4 ("very much"), and the total raw score ranges from 9 to 36. The raw scores will be linearly transformed to a 0 to 100 scale (higher scores represent worse CIPN severity).

SECONDARY OUTCOMES:
Motor Neuropathy at 8 weeks | At 8 weeks
  The 8-item EORTC QLQ-CIPN20 motor subscale will be used to measure motor neuropathy. Each item is rated on a scale from 1 ("not at all") to 4 ("very much"), and the total raw score ranges from 8 to 32. The raw scores will be linearly transformed to a 0 to 100 scale (higher scores represent worse CIPN severity).
Autonomic Neuropathy at 8 weeks | At 8 weeks
  The 3-item EORTC QLQ-CIPN20 autonomic subscale will be used to measure autonomic neuropathy. Each item is rated on a scale from 1 ("not at all") to 4 ("very much"), and the total raw score ranges from 3 to 12. The raw scores will be linearly transformed to a 0 to 100 scale (higher scores represent worse CIPN severity).
Oxaliplatin dose at 8 weeks | At 8 weeks
  Cumulative oxaliplatin dose (mg/m2 of oxaliplatin received) data will be gathered from the electronic medical record (EMR).
Quality of life at 8 weeks | At 8 weeks
  The EORTC QLQ 30-Item Questionnaire (EORTC QLQ-C30) is a patient-reported measure of cancer-specific QOL. Participants rate the degree that each item has applied to them during the past week on a four-point Likert scale (1, not at all; 4, very much). The average of the item scores gives a raw score and the raw score will be transformed to a 0 to 100 scale. Higher scores indicate higher QOL.
Mood at 8 weeks | At 8 weeks
  The 4-item emotional functioning (EF) subscale of the EORTC QLQ-C30 will be used to measure mood. Participants rate the degree that each item has applied to them during the past week on a four-point Likert scale (1, not at all; 4, very much). The average of the item scores gives a raw score and the raw score will be transformed to a 0 to 100 scale. Higher scores indicate improved mood.

OTHER OUTCOMES:
Exercise Adherence - Weekly Minutes of Moderate to Vigorous Physical Activity (MVPA) | Week 1 to week 8
  A heart rate-enabled pedometer will be used to objectively measure adherence in the experimental group. The mean "active minutes" (minutes of moderate-vigorous physical activity) over eight weeks will be collected from a web-based application synchronized with the pedometer.
Total Daily Minutes of MVPA at 8 weeks | At 8 weeks
  The ActiGraph GT3X--a blinded wrist or hip-worn triaxial accelerometer--will be used to objectively measure activity counts per minute. The counts per minute will be transformed to total daily minutes of MVPA.
Adapted Acceptability E-scale | 8 weeks
  The Acceptability E-Scale was adapted to assess acceptability of the walking intervention. Specifically, the survey asks participants to rate the difficulty, enjoyability, helpfulness in managing OIPN symptoms, and acceptability of the time requirement of the MI-Walk intervention. Each item is rated on a scale from one to five and the 15-item survey score ranges from 19 to 75.
Adverse event incidence | Week 1 to week 8
  Intervention-related adverse event incidence will be monitored throughout the study, using brief semi-scripted telephone interviews.
Motivational Interviewing (MI) Fidelity Measure at Study Initiation | Day 1
  An external MI expert will formally review the fidelity of an MI session, using established MI evaluation criteria (the Motivational Interviewing Treatment Integrity Code [MITI]).
MI Fidelity Measure Mid-Study | 6 months
  An external MI expert will formally review the fidelity of an MI session, using the MITI.
MI Fidelity Measure at 9 months | 12 months
  An external MI expert will formally review the fidelity of an MI session, using the MITI.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Kanzawa-Lee, BSN, RN, Principal Investigator — University of Michigan School of Nursing; Ellen M Lavoie Smith, PhD, Principal Investigator — University of Michigan School of Nursing
Locations (7):
- United States (7):
  - The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - St. Joseph Mercy Brighton Health Center, Brighton, Michigan
  - Brighton Center for Specialty Care, Brighton, Michigan
  - St. Joseph Mercy Health System, Canton, Michigan
  - St. Joseph Mercy Chelsea Cancer Center, Chelsea, Michigan
  - The University of Michigan Northville Health Center, Northville, Michigan

REFERENCES:
- [Derived] Kanzawa-Lee GA, Larson JL, Resnicow K, Ploutz-Snyder R, Krauss JC, Smith EML. Home-based aerobic exercise feasibility in oxaliplatin-receiving newly-diagnosed cancer survivors. Eur J Oncol Nurs. 2024 Aug;71:102649. doi: 10.1016/j.ejon.2024.102649. Epub 2024 Jun 27. PMID 38954929